CLINICAL TRIAL: NCT04246606
Title: Retrospective Study Assessing the Concordance of the IHC4 Score Performed in Local Pathology Laboratory or in a Central Laboratory to a Molecular Gold Standard Test Endopredict in Breast Cancer Infiltrating ER+ HER2-
Brief Title: Concordance of the IHC4 Score Performed in Local or Central Laboratory to Endopredict in ER+/HER2- Breast Cancer
Acronym: GEFPICS IHC4
Status: Completed | Type: Observational
Sponsor: UNICANCER (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TRA05-GEFPICS
Record Dates: First submitted 2020-01-23; First posted 2020-01-29 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasm Female
Keywords: IHC4; IHC4+C; Endopredict

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Immunostaining slides for ER, PR, Ki67 and HER2 carry out on surgical resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ER+/HER2- infiltrating early breast cancer: Patients with ER+/HER2- infiltrating early breast cancer for which EndoPredict molecular signature was performed.
  Interventions: Diagnostic Test: IHC4 score

INTERVENTIONS:
Diagnostic Test: IHC4 score — The IHC4 score is a prognostic tool that incorporates immunohistochemical parameters of ER (H-score), PR (% of positive cells), HER2 (positive or negative status), and Ki67 (% of positive cells).
  IHC4 score, combined with nodal status and tumor grade, age, and the type of endocrine therapy (tamoxifen or aromatase inhibitors) provides a clinical score IHC4+C.
  IHC4+C provides a prognostic risk of distant recurrence at 10 years for patients who underwent endocrine therapy for 5 years. IHC4+C defined three distinct risk categories:
  * <10%: low risk
  * [10-20%]: intermediate risk
  * >20%: high risk

SUMMARY:
Retrospective observational, multicentric study assessing the immunohistochemistry (IHC) based test IHC4 score in infiltrating early breast cancer: comparison of the score performed in local laboratory vs in a central laboratory and concordance with a molecular gold standard classifier (EndoPredict).

DETAILED DESCRIPTION:
The IHC4 prognostic signature is an algorithm based on a combination of biomarkers evaluated in immunohistochemistry and anatomical-clinical parameters. Immunohistochemistry is routinely performed as a diagnostic procedure for estrogen receptor (ER; H-score 0-300), progesterone receptor (PR; % of marked cells), HER2 (positive vs negative status) and Ki67 (% of marked cells evaluated by counting). Clinical parameters include lymph node status (0N+, 1-3N+, >3N+, >3N+), tumour size in mm (≤10mm, 11-20, 21-50, >50mm), histologic grade (1, 2, 3), patient's age at diagnosis (<65 years, ≥65 years), and type of treatment (anti-estrogen or aromatase inhibitors).

The method for reading and scoring conditions is very precise and currently guarantee the validity of the test (validated centrally in TransATAC). However, there is not yet an open access web platform available for the calculation of the IHC4 score, due to the prior need for homogenisation of the interpretation of immunochemistry (standardisation of the protocol) to generate a reliable and validated IHC4 under decentralised "real life" conditions. There is currently few published data on the weight of technical parameters (antibody clones, automaton type, etc.) or interpretation methods (scoring) in the calculation of the IHC4 score (IHC4 robustness). However, only one study, published recently, shows a good tolerance of the test to variations in technical protocol or reading.

In this context, a study coordinated by the GEFPICS group, composed of expert pathologists in breast cancer, has been set up to better define the robustness and the scope of IHC4 score. These project will assess 2 main aspects: (i) validate the local "real life" technique for the calculation of the IHC4 score; and (ii) homogenise the IHC reading method (especially for Ki67), on a cohort of cases from the GEFPICS, tested in a prognostic molecular signatures.

ELIGIBILITY:
Sample selection criteria:

1. Prior information of the patient.
2. Histologically proven invasive breast cancer,
3. ER-positive breast cancer, according to the following criteria: ER ≥10 % (local assessment)
4. HER2-negative tumor by IHC (score 0 or 1+) and/or fluorescent in situ hybridization (FISH)/chromogenic in situ hybridization (CISH) negative (local assessment)
5. IHC staining slides for ER, PR, KI67 and HER2 carry out on surgical resection according to local protocol available,
6. In situ hybridization (ISH) staining for HER2 carry out on surgical resection, in case of IHC 2+ for HER2 immunostaining
7. EndoPredict test results available (EPclin),
8. Formalin-fixed and paraffin-embedded (FFPE) block from surgical resection of the primary tumor available,
9. Patient ≥18 years old.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ER+/HER2- infiltrating early breast cancer for which EndoPredict molecular signature was performed.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
To assess the reproducibility of the IHC4 score testing performed in local pathology laboratory (i.e. real life) to in a central laboratory. | Day 1
  Inter-laboratory concordance rate of IHC4 score performed in a local laboratory versus central laboratory. The equivalence of the two methods is defined as a ≥90% concordance rate.

SECONDARY OUTCOMES:
To assess the inter-observer reproducibility of IHC4 scoring carry out by different local pathologists on digitalised slides. | Day 1
  Inter-observer reproducibility of IHC4 scoring carry out by different local pathologists on digitalised slides.
Reproducibility of IHC4+C score compare to the molecular gold standard EPclin (Endopredict). | Day 1
  To assess the consistency of IHC4+C score (IHC4 combined with nodal status and tumor grade) to the molecular gold standard EPclin (Endopredict).
To assess the consistency of the IHC4 scoring performed by a pathologist to an automatic image recognition algorithm. | Day 1
  Inter-observer reproducibility of IHC4 scoring carry out by a pathologist to an automatic image recognition algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Haudebourg, MD, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided